CLINICAL TRIAL: NCT04363580
Title: Creation of Auditory Processing Disorder Screening Tool in French
Acronym: Dépistage TTA
Status: Terminated | Type: Observational
Why Stopped: Inconclusive results
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190844; 2019-A01288-49 (Other: ID RCB)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2023-03

CONDITIONS: Auditory Processing Disorder
Keywords: Auditory processing disorder; Screening tool; Children
MeSH Terms: conditions — Auditory Perceptual Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Children consulting for an assessment of central auditory skills
  Interventions: Other: Auditory processing disorder screening tool

INTERVENTIONS:
Other: Auditory processing disorder screening tool — Screening tool : a questionnaire completed by the parents and the child's teacher and a mini-battery of tests composed of verbal and nonverbal assessments.
  Questions for parents are grouped into four sections:
  * Reference pattern and portrait of the child.
  * Auditory history.
  * History of speech and language development.
  * School history.
  The teacher questionnaire has seven sections:
  * Portrait of the child.
  * Reading and writing.
  * Speaking.
  * Mathematics.
  * Music.
  * Memory.
  * Listening skills and understanding:
    * Concentration and organization.
    * Environment.
  Mini-battery of tests:
  * Dichotic Numeric Listening Test.
  * Identification test of 15 patterns of frequency-varying sounds at each ear.
  * Test of 10 monosyllables in noise per ear.
  * Auditory memory test by measuring the range of figures (instead of words in order to reduce the contribution of language processing).

SUMMARY:
The objective of the study is to validate a screening tool for auditory processing disorder in children of 7 to 13 years old. This screening tool was created based on literature and combines a questionnaire and a mini-battery of tests composed of verbal and nonverbal assessments.

DETAILED DESCRIPTION:
Hearing plays a vital role in the development of a child. Hearing is based on two main systems: the peripheral system and the central system. Peripheral hearing, which includes the outer, middle, and inner ear and the auditory nerve, can detect sound signals.

For its part, the central system, which is composed of auditory structures from the auditory nerve to the brain, makes it possible to process these sound signals and to analyze them. Peripheral hearing damage will result in deafness while a problem in the central auditory system will be called auditory processing disorder. Peripheral deafness can be detected from birth through neonatal screening for deafness. The symptoms of an auditory processing disorder can easily be confused with those caused by attention deficit disorder with or without hyperactivity and a specific language disorder. Auditory processing disorder is often unknown in the medical and educational worlds, and children are referred late for consultation. In addition, the lack of French screening tests for auditory processing disorder and the long waiting lists for specialized consultations help to delay diagnosis and hinder early intervention. Auditory processing disorder affects about 2 to 3% of school-aged children.

The objective of the study is to validate a screening tool for auditory processing disorder in children of 7 to 13 years old. This screening tool was created based on literature and combines a questionnaire and a mini-battery of tests composed of verbal and nonverbal assessments.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 7 to 13 on the day of enrollment.
* Child referred for assessment of central auditory skills, who did not have an auditory processing disorder -type assessment before.
* Hearing thresholds at both ears between 0 decibels Hearing Level (dB HL) and 15 dB HL at 250, 500, 1000, 2000, 4000 and 8000 Hz. Absence of auditory neuropathy.
* Child affiliated to a social security scheme.
* Holders of parental authority who do not oppose the patient's participation in research.

Exclusion Criteria:

* Known neurological disorder (epilepsy, cranial trauma, etc.).
* Non medicated attention deficit since the presence of such a deficit can affect the child's performance during the auditory processing disorder assessment.
* Intellectual disability since impairment of cognitive skills may also explain poor test performance (IQ <80).

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children referred for an assessment of central auditory skills at ENT unit of Necker hospital.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  Comparison of the results of the auditory processing disorder screening tool with those obtained at the auditory processing disorder reference diagnostic battery.
  Sensitivity: Number of true positives / Number of true positives + Number of false negatives
  For the screening tool questionnaire, a score of 1 is given for each item for which parents or teachers believe that the child has a problem. A score of more than 50% on the questionnaire (or sub-section) suggests that the child is at risk of having an auditory processing disorder. The child would also be at risk when he fails at least one hearing test of the tool.
Specificity | 2 years
  Comparison of the results of the auditory processing disorder screening tool with those obtained at the auditory processing disorder reference diagnostic battery.
  Specificity: Number of true negatives / Number of true negatives + Number of false positives
  For the screening tool questionnaire, a score of 1 is given for each item for which parents or teachers believe that the child has a problem. A score of more than 50% on the questionnaire (or sub-section) suggests that the child is at risk of having an auditory processing disorder. The child would also be at risk when he fails at least one hearing test of the tool.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Loundon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Isabelle Rouillon, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No